CLINICAL TRIAL: NCT05738590
Title: Neurophysiological, Sonographical and Pathological Findings in Patients With Inflammatory Versus Degenerative Muscle Diseases
Brief Title: Inflammatory and Degenerative Muscle Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Huda Mahmoud Sayed Abdelal, Resident, Assiut University
Other Study IDs: muscle disease neurophysiology
Record Dates: First submitted 2023-01-24; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Muscle Disease
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- inflammatory muscle disease
  Interventions: Procedure: muscle biopsy
- degenerative muscle disease
  Interventions: Procedure: muscle biopsy

INTERVENTIONS:
Procedure: muscle biopsy — true cut needle biopsy
  Other Names: neurophysiology(nerve conduction,electromyography); muscle ultrasound

SUMMARY:
Correlation between clinical , ultrasonographical, neurophysiological and histopathological findings in muscle diseases of different etiologies.

ELIGIBILITY:
Inclusion Criteria:

1. Muscle diseases of different etiologies.
2. Any age.

Exclusion Criteria:

1. Patient refuse to participate.
2. The anatomy is altered due to severe trauma, tumor , or surgery.
3. Severe deformity preventing examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with muscle disease of different etiologies aged from 18 years to 75 years, of both sex
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
microscopic picture of muscle in inflammatory and degenerative muscle disease | 1 year
  true cut needle muscle biopsy is done to differentiate between inflammatory and degenerative muscle disease in microsopic picture

SECONDARY OUTCOMES:
muscle ultrasound in inflammatory and degenerative muscle disease | 1 year
  muscle ultrasound picture and dimensions in inflammatory and degenerative muscle disease
neurophysiology in inflammatory and degenerative muscle disease | 1 year
  electromyography changes in inflammatory and degenerative muscle disease